CLINICAL TRIAL: NCT06876246
Title: A Digital Health Technology to Prevent Family Violence and Improve Child Mental Health
Brief Title: SBIR/ STTR Family Check-up Online
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY 00001307; R42MH132191 (NIH)
Record Dates: First submitted 2025-02-11; First posted 2025-03-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Mental Health; Parenting Stress; Academic Achievement; Parenting Skills; Behavior Problems
Keywords: digital health; implementation science; mental health; family intervention; school-based intervention
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FCU Online with telehealth coaching (Experimental): FCU Online Digital intervention with telehealth coaching. This arm includes usage of the digital intervention plus telehealth support from a parenting coach.
  Interventions: Behavioral: FCU Online with Telehealth Coaching
- FCU Online (Experimental): FCU Online digital intervention. This arm includes use of the digital intervention only (i.e., no telehealth coaching).
  Interventions: Behavioral: Family Check-Up Online
- Providers participating in feasibility/ acceptability interviews (No Intervention): School-based providers will be interviewed to help the research team identify feasible and acceptable implementation strategies for delivery of the basic and supported FCU Online models as routine school services.
- Parents participating in feasibility/ acceptability interviews (No Intervention): Parents of middle school-aged students will be interviewed to help the research team identify feasible and acceptable implementation strategies for delivery of the basic and supported FCU Online models as routine school services.

INTERVENTIONS:
Behavioral: Family Check-Up Online — The Family Check-Up Online is a digital intervention that includes an assessment, computer-generated feedback, and intervention modules that focus on improving family relationships and parenting skills in order to reduce child mental health problems and to improve child self-regulation. These modules include Healthy Behaviors for Stressful Times, Positive Parenting, Rules and Consequences, Supporting School Success, and Communication.
  Arms: FCU Online
Behavioral: FCU Online with Telehealth Coaching — This intervention is the Family Check-Up Online plus telehealth support from a parenting coach. The Family Check-Up Online is a digital intervention that includes an assessment, computer-generated feedback, and intervention modules that focus on improving family relationships and parenting skills in order to reduce child mental health problems and to improve child self-regulation. These modules include Healthy Behaviors for Stressful Times, Positive Parenting, Rules and Consequences, Supporting School Success, and Communication. A coach based at the child's school meets with caregivers via telehealth modality to provide motivation and to help caregivers tailor the content of the modules to their specific child and family's needs.
  Arms: FCU Online with telehealth coaching

SUMMARY:
The Family Check-Up Online, a digital health intervention, was designed to improve child mental health through family-centered intervention. The Family Check-Up is grounded in over 25 years of evidence-based research and has been shown to improve child mental health and behavior including depression and conduct problems. The investigators were supported by an SBIR Phase I award (R43MH132191) to evaluate the feasibility and acceptability of the digital health product in schools and to adapt the product based on findings of that work. Findings from that project suggested the model is a good fit for schools, with school providers stating a need for family-centered interventions that target child behavior and mental health, but with few resources or evidence-based programs available. The research team received feedback that suggests the model should be evaluated as both an uncoached version and coached version, delivered with provider support. In the current project, the investigators plan to continue work in schools to develop the model for commercialization, including understanding the process for embedding the FCU Online into current student support systems and implementation factors that lead to maintenance of the model in schools. The investigators plan to conduct a hybrid type 2 effectiveness-implementation trial to evaluate the effectiveness of the FCU Online when delivered by real world providers. Thirty providers (N=600 students/families) will be randomly assigned to receive training in the FCU Online coached vs. uncoached models. The research team will then evaluate outcomes including family relationships, parenting skills, and child mental health and behavior. The investigators predict that the FCU Online will improve child mental health and behavior, and will test for moderators such as provider training and child baseline risk. Findings will have implications for commercialization of the product in schools and implementation of the model in a range of different school settings.

DETAILED DESCRIPTION:
In this study the investigators propose the following specific aims:

1. Examine the feasibility and acceptability of embedding the FCU Online model into multi-tiered systems of support (MTSS). The investigative team (comprised of researchers and school partners) will (1a) identify strategies to reach students at risk for poor mental health outcomes using natural indicators within the school environment. Then, the team will (1b) identify feasible and acceptable implementation strategies for delivery of the basic (i.e., no coaching) and supported (i.e., with coaching) FCU Online models as routine school services. Phase 1 data suggest that schools vary in their preference for a coached vs. uncoached delivery system. The investigators will explore the best strategies for delivery of both models in a series of interviews with N=20 school providers and N=20 parents that will guide the Aim 2 effectiveness trial.
2. Conduct a comparative effectiveness trial to examine outcomes associated with the FCU Online model in school delivery systems. The investigators will examine the effectiveness of the FCU Online for middle school youth in a hybrid type 2 effectiveness-implementation trial. Based on Phase 1 results, 30 school providers across multiple districts will be randomly assigned to deliver the basic (i.e., no coaching) or supported (i.e., with coaching) digital health model. Each provider will enroll 20 families/students (N=600) in the intervention across one year. The investigators will test parent and student outcomes associated with the program over a 6-month period including student mental health and behavior problems. Potential moderators of family engagement and improved outcomes, including pre-existing risk (family and student level) and provider characteristics, will be examined. The investigators hypothesize greater effects of The FCU Online with coaching for students with high baseline behavior problems and for providers with experience working with high-risk students. Moderation analysis results will highlight which students might benefit most from the FCU Online with coaching and from which providers.
3. Examine factors related to successful implementation in schools that will guide future commercialization. Guided by the RE-AIM implementation framework, the investigators will evaluate factors related to Reach (percent of students who received FCU Online supports), Adoption (who engages at schools and to what extent), Implementation (fidelity monitoring and usage),and Maintenance (provider usage at end of clinical trial) of the FCU Online models. These analyses will inform commercialization and funding models for the product in school delivery systems and future plans for Phase III funding.

ELIGIBILITY:
Inclusion Criteria:

* A caregiver must have a child between the ages of 11 and 14 enrolled at a participating school;
* the caregiver must be the parent or legal guardian of the youth;
* the caregiver must have a smartphone with text messaging capability and access to email; and
* the youth must be identified by school providers as needing or being eligible for Tier 2 or Tier 3 supports or services.

Exclusion Criteria:

* the caregiver is unable to read in either English or Spanish; or
* the family is already participating in another study of the University of Oregon's Prevention Science Institute.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1270 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Child Depression (Parent report) | baseline, 6 months
  Parents report on their child's depression using the two item PHQ-2. Scores for the individual items range from 0 (not at all) to 3 (nearly all) and are summed together. Higher scores indicate greater child depression.
Change from Baseline in Child Anxiety (Parent report) | baseline, 6 months
  Parents report on their child's anxiety using the two item GAD-2. Scores for the individual items range from 0 (not at all) to 3 (nearly all) and are summed together. Higher scores indicate greater child anxiety.
Change from Baseline in Positive Parenting (Parent report) | baseline, 6 months
  Parents report on their use of positive parenting skills using a modified version of the Parenting Young Children scale. Parents are asked to indicate the frequency with which they used positive parenting skills (such as encouragement and praise, relationship building, giving clear directions, and using rewards for positive behavior) over the past month using a 5-pt scale (0=Never/ 1=Rarely/ 2= Sometimes/ 3=Often/ 4=Very Often). Responses to these 10 items are summed. Higher scores indicate frequent use of positive parenting skills.
Change from Baseline in Rules and Consequences (Parent report) | baseline, 6 months
  Parents report on the extent to which they enforced rules and consequences for negative behavior over the past month using a 13-item scale developed for this project. Parents are asked to indicate the frequency with which they monitored their child's behavior, set clear rules, applied logical consequences, and ignored annoying behavior using a 5-pt scale (0=Never/ 1=Rarely/ 2= Sometimes/ 3=Often/ 4=Very Often). Responses are summed and higher scores indicate more consistent use of rules and consequences.
Change from Baseline in Positive Communication (Parent report) | baseline, 6 months
  Parents report on the extent to which positive communication occurred with their child over the past month using a 12-item scale developed for this project. Parents are asked to indicate the frequency with which they communicated calmly and clearly, listened to their child, and mitigated conflict using a 5-pt scale (0=Never/ 1=Rarely/ 2= Sometimes/ 3=Often/ 4=Very Often). Responses are summed and higher scores indicate more positive communication within the family.
Change from Baseline in Supporting School Success (Parent report) | baseline, 6 months
  Parents report on the ways they support their child's school success over the past month using a16-item scale developed for this project. Parents are asked to indicate the frequency with which their family followed regular morning, meal, sleep, school, and homework routines using a 5-pt scale (0=Never/ 1=Almost Never/ 2= Sometimes/ 3=Frequently/ 4=Almost Always). Responses are summed, and higher scores indicate more frequent use of routines that support school success.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Mauricio, PhD, Principal Investigator — University of Oregon; Lisa A Reiter, PhD, Principal Investigator — Northwest Prevention Science; Elizabeth A Stormshak, PhD, Principal Investigator — Northwest Prevention Science
Locations (1):
- Prevention Science Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
External researchers will have access to de-identified, individual-level data, and members of the general public will have access to metadata, descriptive data, and summary data. External researcher requests for individual-level data must be accompanied by a signed Data Use Agreement, and researchers must document that they are working under an institution with a Federal Wide Assurance (FWA). University of Oregon Information Services staff will develop and maintain the enclave to host and provide access to de-identified study data. The data enclave will be accessible to qualified researchers through a web portal that has capabilities to send and receive data by using encrypted secure transmission protocols.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual-level data will be released 12 months after the final participant has completed a given wave of data collection. This will allow time for data cleaning, and also provides a brief window for the investigative team to analyze and publish key findings prior to sharing the data, but still makes the data available to external researchers in a timely manner. After the grant award ends, if no additional external support is available to provide access to the data, the investigators will partner with the University of Oregon Libraries to host the data enclave and provide access to the data in perpetuity.
Access Criteria: External researcher requests for de-identified individual-level data must be accompanied by a signed Data Use Agreement, and researchers must document that they are working under an institution with a Federal Wide Assurance (FWA).To optimize usage of the data, the website at Northwest Prevention Science, Inc. will provide clear instructions for accessing the data.
URL: https://www.nwpreventionscience.org/